CLINICAL TRIAL: NCT05578703
Title: Gastric Fundus Ablation Plus Endoscopic Sleeve Gastroplasty for Weight Loss
Brief Title: ABLATE WEIGHT (Ablation Plus ESG for Weight Loss)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: True You Weight Loss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-001
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gastric Fundic Ablation plus Endoscopic Sleeve Gastroplasty (Experimental): Subjects will undergo fundic mucosal ablation followed by endoscopic sleeve gastroplasty
  Interventions: Procedure: Fundic Ablation Sequentially in Combination with Endoscopic Sleeve Gastroplasty; Device: Fundic Mucosal Ablation with ERBE HybridAPC; Device: Apollo ESG

INTERVENTIONS:
Procedure: Fundic Ablation Sequentially in Combination with Endoscopic Sleeve Gastroplasty — Fundic mucosal ablation followed by endoscopic sleeve gastroplasty in the treatment of adults with obesity
Device: Fundic Mucosal Ablation with ERBE HybridAPC — Fundic mucosal ablation utilizing approved ERBE HybridAPC
Device: Apollo ESG — Using only Apollo ESG as approved per label

SUMMARY:
The purpose of this research is to investigate the effects of fundic ablation (FA) on circulating plasma ghrelin, satiation, and total body weight loss, as well as the incidence of adverse events. This procedure will be carried out with the HybridAPC (ERBE Elektromedizin GmbH, Tübingen, Germany). The HybridAPC instrument creates an electric current to deliver a safe amount of thermal injury to a portion of the stomach known as the gastric fundus. This thermal injury will target a hormone called ghrelin which is the only known hormone linked to increasing appetite, calorie intake, and weight gain. This procedure is designed to target the bodily effects of appetite control and gastric sensory and motor functions which cause the feeling of fullness and satiation. The fundic mucosal ablation is not typically done prior to the endoscopic sleeve gastroplasty procedure. When fundic mucosal ablation is sequentially paired with endoscopic sleeve gastroplasty (ESG), this combined investigational approach may lead to decreased fasting ghrelin levels, improved satiation, and greater total body weight loss than traditional ESG. This study will help determine if the combined impact of FA with ESG should be made available to patients as part of a comprehensive weight loss strategy.

DETAILED DESCRIPTION:
Obesity is a chronic disease state driven by the imbalance of caloric intake and expenditure and mediated by multiple central and peripheral pathways that may serve as targets for therapeutic interventions. The endoscopic sleeve gastroplasty (ESG) is a per oral gastric remodeling technique that employs full-thickness suturing to imbricate the stomach along the greater curvature to achieve a restricted, sleeve-like configuration. While the ESG recapitulates the configuration of a gastric sleeve, it has not yet been shown to achieve as robust weight loss outcomes compared to the laparoscopic sleeve gastrectomy (LSG). A major difference between ESG and LSG is that the former does not involve the gastric fundus. The proximal stomach, and the fundus in particular, produces ghrelin, the only known orexigenic hormone, which has been linked to increased calorie intake and weight gain. Studies have observed reduced levels of ghrelin along multiple timepoints following LSG, and this has been attributed to targeting of the fundus, as bariatric surgeries that did not involve the fundus did not see a decrease in circulating plasma ghrelin. In contrast, in a small comparative study of ESG and LSG, patients who had undergone ESG did not show any decrease in fasting ghrelin levels, 8 ostensibly due to fundic-sparing. In this study, the investigators propose to investigate the effects of fundic ablation (FA) on circulating plasma ghrelin, satiation via standard nutrient drink test, and total body weight loss (TBWL), as well as the incidence of adverse events. Fundic ablation will be followed sequentially with ESG, to evaluate the combined impact of FA and ESG (FA-ESG). This study hypothesizes that, compared to baseline, FA-ESG will diminish fasting ghrelin levels, improve satiation, and induce a TBWL ≥ 15% at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 21-65
2. Body mass Index (BMI) ≥30 kilograms per square meter (kg/m²), or ≤50 kg/m²
3. History of at least one unsuccessful dietary effort to lose body weight
4. Willing and able to participate in the study procedures
5. Understand and voluntarily sign the informed consent
6. Approved ESG candidate at TYWL
7. Access to internet
8. Reliable transportation to and from Cary, North Carolina surrounding area

Exclusion Criteria:

1. Younger than 21 years of age
2. Older than 65 years of age
3. Patients on any medications or supplements including those that may influence cholecystokinin (CCK), glucose, growth hormone, insulin and/or somatostatin levels
4. Milk and/or soy allergies
5. History of any stomach manipulation (including repair of hiatal hernia)
6. History of disordered eating
7. Patients who do not give their consent to the enrollment in the study or are incompetent, unconscious or unable to express their consent for any reason
8. Hemoglobin A1c > 7.0 or any patient with symptoms suggestive of gastroparesis or a formal diagnosis of gastroparesis
9. Patients taking the following medications known to impair gastric accommodation: buspirone, mirtazapine
10. Patients taking the following medications known to accelerate or impair gastric emptying: Reglan (metoclopramide), Zelnorm (tegaserod), Motegrity (prucalopride), erythromycin, Motilium (domperidone), opiates, anticholinergic agents
11. Patients who are pregnant or who plan to become pregnant during study duration
12. Use of non-steroidal anti-inflammatory medications without the ability to stop these during study duration
13. Patients on chronic anticoagulation
14. History of functional gastrointestinal disorder, including functional dyspepsia, irritable bowel syndrome, or other syndromes known to affect gastric sensorimotor function.
15. Concurrent use of weight loss medications.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Fasting Plasma Ghrelin Levels | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, and Month 18
  Change from baseline for the quantitative determination of fasting ghrelin, total plasma measured by EIA/ELISA laboratory assays
Change from Baseline in Timed Standardized Nutrient Drink Test | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, and Month 18
  Measure timed consumption of a standardized nutrient drink test utilizing a sensation of satiation visual analogue scale. The severity of symptoms range from 0 (no symptoms) to 5 (maximum or unbearable fullness/satiation) and will measure volume to comfortable fullness (VTF) and maximum tolerated volume (MTV)
Change from Baseline in Gastroparesis Cardinal Symptom Index (GCSI) | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, and Month 18
  Assess the severity of patient-reported gastroparesis symptoms. The GCSI gastroparesis symptoms score ranges from 0-none to 5-very severe. High scores reflect greater symptom severity
Change from Baseline in Daily Eats: Measuring Daily Eating Factors (DAILY EATS) | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, and Month 18
  Rate the responses to the DAILY EATS questionnaire. The DAILY EATS questionnaire is designed to better understand patient's definitions, experience, and importance, of eating-related factors on a scale of 0-10. The DAILY EATS is a 5-item, patient-reported measure evaluating key eating-related factors (Worst and Average Hunger, Appetite, Cravings, and Satiety)
Percent Change in Total Body Weight Loss (TBWL) from Baseline | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 14, Month 15, Month 16, Month 17, and Month 18
  Measure percent change in total body weight over time following FA alone and FA-ESG. TBWL = pre-op weight - post op body weight. % TBWL is the fraction of body weight expressed in percentage term
Change from Baseline in Weight Efficacy Life-Style Questionnaire Short Form (WEL-SF) composite score | Baseline, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, and Month 18
  Measure of eating self-efficacy consisting of 8-items on a scale of 0 (not at all confident) to 10 (very confident)

SECONDARY OUTCOMES:
Rate of safety and adverse events | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 14, Month 15, Month 16, Month 17, and Month 18
  FA and FA-ESG safety will be measured by the rate of serious adverse events (SAEs), adverse events (AEs), and accommodative symptom occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E McGowan, MD, MSCR, Principal Investigator — CEO/ Medical Director
Locations (1):
- True You Weight Loss, Cary, North Carolina, United States

REFERENCES:
- [Background] Fukunishi Y. [Electron microscopic findings in peripheral nerve lesions of nude mouse inoculated with M. leprae--perineural lesion]. Nihon Rai Gakkai Zasshi. 1985 Jul-Sep;54(3):82-7. doi: 10.5025/hansen1977.54.82. No abstract available. Japanese. PMID 3915747
- [Background] Cummings DE, Overduin J. Gastrointestinal regulation of food intake. J Clin Invest. 2007 Jan;117(1):13-23. doi: 10.1172/JCI30227. PMID 17200702
- [Background] Goitein D, Lederfein D, Tzioni R, Berkenstadt H, Venturero M, Rubin M. Mapping of ghrelin gene expression and cell distribution in the stomach of morbidly obese patients--a possible guide for efficient sleeve gastrectomy construction. Obes Surg. 2012 Apr;22(4):617-22. doi: 10.1007/s11695-011-0585-9. PMID 22231739
- [Background] Anderson B, Switzer NJ, Almamar A, Shi X, Birch DW, Karmali S. The impact of laparoscopic sleeve gastrectomy on plasma ghrelin levels: a systematic review. Obes Surg. 2013 Sep;23(9):1476-80. doi: 10.1007/s11695-013-0999-7. PMID 23794092
- [Background] McCarty TR, Jirapinyo P, Thompson CC. Effect of Sleeve Gastrectomy on Ghrelin, GLP-1, PYY, and GIP Gut Hormones: A Systematic Review and Meta-analysis. Ann Surg. 2020 Jul;272(1):72-80. doi: 10.1097/SLA.0000000000003614. PMID 31592891
- [Background] Langer FB, Reza Hoda MA, Bohdjalian A, Felberbauer FX, Zacherl J, Wenzl E, Schindler K, Luger A, Ludvik B, Prager G. Sleeve gastrectomy and gastric banding: effects on plasma ghrelin levels. Obes Surg. 2005 Aug;15(7):1024-9. doi: 10.1381/0960892054621125. PMID 16105401
- [Background] Lopez-Nava G, Negi A, Bautista-Castano I, Rubio MA, Asokkumar R. Gut and Metabolic Hormones Changes After Endoscopic Sleeve Gastroplasty (ESG) Vs. Laparoscopic Sleeve Gastrectomy (LSG). Obes Surg. 2020 Jul;30(7):2642-2651. doi: 10.1007/s11695-020-04541-0. PMID 32193741
- [Background] Vijayvargiya P, Chedid V, Wang XJ, Atieh J, Maselli D, Burton DD, Clark MM, Acosta A, Camilleri M. Associations of gastric volumes, ingestive behavior, calorie and volume intake, and fullness in obesity. Am J Physiol Gastrointest Liver Physiol. 2020 Aug 1;319(2):G238-G244. doi: 10.1152/ajpgi.00140.2020. Epub 2020 Jul 6. PMID 32628074
- [Background] Fayad L, Oberbach A, Schweitzer M, Askin F, Voltaggio L, Larman T, Enderle M, Hahn H, Khashab MA, Kalloo AN, Kumbhari V. Gastric mucosal devitalization (GMD): translation to a novel endoscopic metabolic therapy. Endosc Int Open. 2019 Dec;7(12):E1640-E1645. doi: 10.1055/a-0957-3067. Epub 2019 Nov 25. PMID 31788546
- [Background] Chial HJ, Camilleri C, Delgado-Aros S, Burton D, Thomforde G, Ferber I, Camilleri M. A nutrient drink test to assess maximum tolerated volume and postprandial symptoms: effects of gender, body mass index and age in health. Neurogastroenterol Motil. 2002 Jun;14(3):249-53. doi: 10.1046/j.1365-2982.2002.00326.x. PMID 12061909
- [Background] Lopez Nava G, Arau RT, Asokkumar R, Maselli DB, Rapaka B, Matar R, Bautista I, Espinos Perez JC, Bilbao AM, Jaruvongvanich V, Vargas EJ, Storm AC, Neto MG, Abu Dayyeh BK. Prospective Multicenter Study of the Primary Obesity Surgery Endoluminal (POSE 2.0) Procedure for Treatment of Obesity. Clin Gastroenterol Hepatol. 2023 Jan;21(1):81-89.e4. doi: 10.1016/j.cgh.2022.04.019. Epub 2022 May 6. PMID 35533995
- [Background] Fastenau J, Rozjabek H, Qin S, McLeod L, Nelson L, Ma J, Harris N. Psychometric evaluation of the DAILY EATS questionnaire in individuals living with obesity. J Patient Rep Outcomes. 2020 Nov 23;4(1):99. doi: 10.1186/s41687-020-00259-w. PMID 33226548
- [Background] Ames GE, Heckman MG, Diehl NN, Grothe KB, Clark MM. Further statistical and clinical validity for the Weight Efficacy Lifestyle Questionnaire-Short Form. Eat Behav. 2015 Aug;18:115-9. doi: 10.1016/j.eatbeh.2015.05.003. Epub 2015 May 21. PMID 26042918